CLINICAL TRIAL: NCT03064386
Title: Comparative Study of Postieror Malleolar Fracture With Plate and Screw Fixation
Brief Title: Comparative Study of Postieror Ankle Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Liming Cheng, Professor, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56014768-6
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Postieror Malleolar Fracture; Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plate group (Experimental): internal fixation with the plate
  Interventions: Procedure: Plate fixation
- screw group (Experimental): internal fixation with the screw
  Interventions: Procedure: Screw fixation

INTERVENTIONS:
Procedure: Plate fixation — internal fixation with the plate
  Arms: plate group
Procedure: Screw fixation — internal fixation with the screw
  Arms: screw group

SUMMARY:
To compare the clinical efficacy of open reduction and internal fixation (ORIF) with plate and screw for postieror malleolar fractures.

ELIGIBILITY:
Inclusion Criteria:

supination-external rotation Ⅳ type injury

Exclusion Criteria:

Pion fracture; Isolated posterior ankle fracture.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-28 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
functional score | One year after surgery
  AOFAS function score for ankle